CLINICAL TRIAL: NCT06646575
Title: Exploring the Experience of Patients, Carers, and Healthcare Clinicians of the CGA-Q, a Tool to Facilitate Person-centred Comprehensive Geriatric Assessment (CGA)
Brief Title: Exploring the User Experience of CGA-Q
Status: Completed | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 337803
Record Dates: First submitted 2024-10-08; First posted 2024-10-17 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: CGA; Comprehensive Geriatric Assessment; Person Centred Care; Frailty
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patient participant
  Interventions: Other: Qualitative data, no intervention
- Informal carer participant
  Interventions: Other: Qualitative data, no intervention
- Healthcare professional participant
  Interventions: Other: Qualitative data, no intervention

INTERVENTIONS:
Other: Qualitative data, no intervention — This is a qualitative study

SUMMARY:
* As people become older they may start to have more than one health issue at one time.
* Geriatricians are doctors who specialise in looking after older people.
* A tool that geriatricians use is the Comprehensive Geriatric Assessment (CGA).
* Its purpose is to make sure that all parts of an older person's health are looked after. This includes their physical, psychological, social, environmental, and functional health.
* The problem with CGA is that sometimes it does not focus on what is important to the patient.
* When a clinician makes sure that they are looking after the things that are most important to a patient this is called person-centred care.
* The CGA-Q is a questionnaire. It aims to improve how person-centred someone's care.
* This study aims to find out what people think of CGA-Q.

DETAILED DESCRIPTION:
Comprehensive Geriatric Assessment (CGA) is a multi-disciplinary, multi-domain intervention that involves reviewing an older person's physical, psychological, social and environmental health and then implementing a plan in collaboration with the patient. Its purpose is to facilitate a holistic assessment of an older person that considers the multiple, and potentially overlapping, issues they may be experiencing.

Cochrane reviews have shown that when CGA is delivered in an inpatient setting it reduces the risk of an individual dying or moving into a care facility. It has also been shown, through randomised control trials, to improve outcomes in the perioperative, hospital-at-home, and oncology setting. As a result, it is considered the gold-standard for managing frailty in older adults.

Person-centred care describes care that is focused on the needs and expectations of an individual, rather than a single disease or process. It improves the individual's quality of life and their satisfaction with their care. Its impact on outcomes is such that the World Health Organisation has called for it to be a key priority in healthcare delivery. Person-centred care is heralded as the gold-standard method for delivering care.

Currently, research on person-centred care primarily focuses on how an individual can measure whether care is person-centred. Conversely, there is clinical equipoise in regards to how a clinician can be supported to deliver person-centred CGA. The CGA-Q is a tool that is currently being used as part of routine care in some outpatient CGA clinics in the NHS and it seeks to facilitate person-centred care. The CGA-questionnaire was adapted from the CGA-GOLD questionnaire, which is validated for use in the outpatient older person's oncology service. The CGA-GOLD questionnaire's purpose is to identify which older person needs to undergo a CGA. However, the CGA-questionnaire differs significantly from this as its purpose is not for a needs assessment but instead to facilitate person-centred care. To understand the acceptability and impact of the CGA-Q and how it integrates into an NHS service the investigators will conduct focus groups with stakeholders including patients, carers, and healthcare professionals. The aim is to understand the stakeholder experience of using the CGA-Q. The investigators will also seek to understand the experience of engaging with CGA and their opinions of person-centred care.

By understanding the experience of using the CGA-Q the investigators will be able to generate an evidence base to inform its future use and wider application in healthcare services.

ELIGIBILITY:
Inclusion Criteria:

* Patient inclusion criteria:

  * Age 65 years or older
  * Attending an outpatient CGA appointment
  * Completed a CGA-Q as part of standard care
  * English speaking
  * Have sufficient cognitive function to participate in a focus group
  * Have capacity to consent to participating in the study

Informal carer inclusion criteria:

* Age 18 years or older
* An informal carer for a patient who is attending an outpatient CGA appointment
* An informal carer for a patient who has completed a CGA-Q as part of standard care
* Attending the outpatient appointment with the individual they care for
* The person they care for consents to their informal carers participation in the study
* English speaking
* Have sufficient cognitive function to participate in a focus group
* Have capacity to consent to participating in the study

Healthcare professional inclusion criteria:

* A registered healthcare professional
* Involved in the delivery of an outpatient CGA appointment
* Has been involved in the episode of care during which a patient and or their carer completed the CGA-Q

Exclusion Criteria:

* Patient exclusion criteria:

  * Assessed by the clinical care team to be too clinically unstable to participate in the study
  * Declines to participate
  * Not able to attend the focus group on the pre-set date

Informal carer exclusion criteria:

* Age less than 18 years
* Cares for the patient as part of their employment
* Declines to participate
* Not able to attend the focus group on the pre-set date

Healthcare professional exclusion criteria:

* Not involved in the delivery of an outpatient CGA clinic
* Has not seen any patients who have completed the CGA-Q
* Declines to participate
* Not able to attend the focus group on the pre-set date

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Individuals who have experienced the CGA-Q either as a healthcare professional or as a patient or informal carer of a patient
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2024-11-04 (Actual); Primary Completion 2025-03-17 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Participants experience of the CGA-Q and its impact on person-centred care | 3 months
  This data will consist of qualitative data collected through three separate focus group discussions with patients, informal carers, and health care professionals

CONTACTS AND LOCATIONS:
Locations (1):
- Guy's and St Thomas' NHS Foundation trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Society, B. G. (2019). Comprehensive Geriatric Assessment Toolkit for Primary Care Practitioners. B. G. Society. https://www.bgs.org.uk/sites/default/files/content/resources/files/2019-02-08/BGS%20Toolkit%20-%20FINAL%20FOR%20WEB_0.pdf
- [Background] Ellis G, Gardner M, Tsiachristas A, Langhorne P, Burke O, Harwood RH, Conroy SP, Kircher T, Somme D, Saltvedt I, Wald H, O'Neill D, Robinson D, Shepperd S. Comprehensive geriatric assessment for older adults admitted to hospital. Cochrane Database Syst Rev. 2017 Sep 12;9(9):CD006211. doi: 10.1002/14651858.CD006211.pub3. PMID 28898390
- [Background] Partridge JS, Harari D, Martin FC, Dhesi JK. The impact of pre-operative comprehensive geriatric assessment on postoperative outcomes in older patients undergoing scheduled surgery: a systematic review. Anaesthesia. 2014 Jan;69 Suppl 1:8-16. doi: 10.1111/anae.12494. PMID 24303856
- [Background] Shepperd S, Cradduck-Bamford A, Butler C, Ellis G, Godfrey M, Gray A, Hemsley A, Khanna P, Langhorne P, Makela P, Mort S, Ramsay S, Schiff R, Singh S, Smith S, Stott DJ, Tsiachristas A, Wilkinson A, Yu LM, Young J. Hospital at Home admission avoidance with comprehensive geriatric assessment to maintain living at home for people aged 65 years and over: a RCT. Southampton (UK): NIHR Journals Library; 2022 Jan. Available from http://www.ncbi.nlm.nih.gov/books/NBK577408/ PMID 35129936
- [Background] Soo WK, King MT, Pope A, Parente P, Darzins P, Davis ID. Integrated Geriatric Assessment and Treatment Effectiveness (INTEGERATE) in older people with cancer starting systemic anticancer treatment in Australia: a multicentre, open-label, randomised controlled trial. Lancet Healthy Longev. 2022 Sep;3(9):e617-e627. doi: 10.1016/S2666-7568(22)00169-6. Epub 2022 Aug 22. PMID 36102776
- [Background] World Health Organization, W. (2015). WHO global strategy on people-centred and integrated health services: interim report. https://www.afro.who.int/sites/default/files/2017-07/who-global-strategy-on-pcihs-main-document_final.pdf
- [Background] Poochikian-Sarkissian S, Sidani S, Ferguson-Pare M, Doran D. Examining the relationship between patient-centred care and outcomes. Can J Neurosci Nurs. 2010;32(4):14-21. PMID 21268489
- [Background] Whittle AK, Kalsi T, Babic-Illman G, Wang Y, Fields P, Ross PJ, Maisey NR, Hughes S, Kwan W, Harari D. A comprehensive geriatric assessment screening questionnaire (CGA-GOLD) for older people undergoing treatment for cancer. Eur J Cancer Care (Engl). 2017 Sep;26(5). doi: 10.1111/ecc.12509. Epub 2016 May 1. PMID 27132979